CLINICAL TRIAL: NCT06560372
Title: Incidence, Characteristics and Evolution of Cerebral Vasospasm With Clinical Impact in Moderate to Severe Traumatic Brain Injury Complicated by Subarachnoid Hemorrhage at Martinique University Hospital
Acronym: VASO-TC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23_RIPH2-14
Record Dates: First submitted 2024-07-23; First posted 2024-08-19 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: SAH (Subarachnoid Hemorrhage); Cerebral Vasospasm; Moderate Traumatic Brain Injury; Severe Traumatic Brain Injury
Keywords: SAH (Subarachnoid Hemorrhage); Cerebral Vasospasm; Moderate and severe Traumatic Brain Injury; CT scan; Cerebral perfusion
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Brain Injuries, Traumatic; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Patients hospitalized at Martinique University Hospital for treatment or monitoring of a moderate or severe TBI (Glasgow Score less than or equal to 13 at initial treatment) presenting with SAH on initial cerebral CT scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment or monitoring of a moderate or severe TBI presenting with SAH on initial cerebral CT scan (Experimental): Patients hospitalized at Martinique University Hospital for treatment or monitoring of a moderate or severe TBI (Glasgow Score less than or equal to 13 at initial treatment) presenting with SAH on initial cerebral CT scan.
  Any head trauma patient with an altered level of consciousness must benefit, as part of routine care, from clinical monitoring and a CT imaging assessment, as well as the opinion of the doctor on duty in the resuscitation department.
  If the patient has a traumatic SAH on the cerebral CT scan, he must benefit from an injected sequence exploring the supra-aortic trunks. If there is evidence of intracranial hypertension on cerebral CT or abnormal transcranial doppler, they will benefit, according to the service protocol, from the placement of a parenchymal intracranial pressure sensor. These patients also benefit from clinical monitoring in critical care, as well as a daily biological assessment.
  Interventions: Procedure: Additional realization of a brain perfusion scan sequence which would allow the radiological diagnosis of CV

INTERVENTIONS:
Procedure: Additional realization of a brain perfusion scan sequence which would allow the radiological diagnosis of CV — Neurological monitoring by daily TCD will be carried out.
  * If monitoring finds, between 3rd and 12th day of treatment, a neurological deterioration or an uncontrolled increase in intracranial pressure, a new cerebral CT scan will be performed, as recommended in such a case.
  * As part of this research, a specific interventional act will be implemented: additional brain perfusion scan sequence which would allow the radiological diagnosis of CV.
  * Interventions related to improving cerebral perfusion and reducing intracranial pressure recommended in head trauma patients will be implemented without modification of management linked to protocol.
  The additional perfusion sequences will be analyzed independently and blindly by 2 experienced interventional neuroradiologists (double reading blinded to the patient's characteristics).

SUMMARY:
Context :

Moderate to severe head trauma with altered state of consciousness is an extremely common pathology (between 60 and 120 cases per 100 000 people per year depending on the country and age group), and is responsible for 30% of deaths by trauma. It is complicated in 30-60% of cases by subarachnoid hemorrhage (SAH), which makes it the leading cause of SAH. SAH and its complications are well described when the origin is aneurysmal, notably cerebral vasospasm (CV) because it promotes delayed cerebral ischemia with a major prognostic impact. This is why the screening and prevention of this vasospasm are well established in the literature and in practice, in the nosological context of aneurysmal SAH.

Research problem :

However, when it comes to post-traumatic SAH, CV is a more maligned entity, with a much less detailed description. However, when we know the prognostic interest that it could have for patients, it seems legitimate to seek to define its physiopathological and epidemiological contours. On a prospective cohort of 290 subjects, Oertel et al. (2005) demonstrated, in head trauma patients, an incidence of approximately 40% of compatible signs with the recognized criteria of CV.

To date, the literature remains sparse on this subject.

Proposed study :

In view of the incomplete scientific literature, the study team wish to carry out a prospective epidemiological study in moderate to severe head trauma patients complicated by SAH and hospitalized at the Martinique University Hospital, with the aim of better characterizing the incidence of the occurrence, and evolution of CV with clinical impact in these patients.

One of the original aspects of the proposed study is the use of CT scan with perfusion sequence, which has shown its superiority to Transcranial Doppler. The other particularity is its prospective aspect and triggered by an alteration in the clinical state of the patient presenting a traumatic SAH, then directly linking the pathophysiology (cerebral ischemia) and the clinical impact. Thus, the diagnosis of traumatic CV will be made on a cerebral CT scan by the association of the 50% reduction in the caliber of one or more cerebral arteries and a perfusion defect in the perfusion sequence in a context of alteration of neurological clinical examination or deterioration of neurological monitoring parameters. Finally, few studies have monitored the evolution of these patients at 1 and 6 months after the initial event.

Hypothesis :

The research hypothesis is that in the population of moderate to severe head trauma patients hospitalized at the Martinique University Hospital, when a new neurological symptomatology or a deterioration in the state of consciousness occurs, it could be a post-truamatic CV in 15 to 20% of cases.

Indeed, the rare studies find frequencies of radiologically confirmed CV in head trauma patients of around 30-45%, with low numbers of subjects, retrospective studies, or not correlated with the clinic and with the clinical and paraclinical data necessary for the positive diagnosis of this entity. The reported frequency of traumatic CV with clinical impact ranges between 15-20%.

The study team therefore expect an incidence of 15 to 20% of CV with clinical impact in patients with traumatic SAH in Martinique. CV could be responsible for sudden deterioration of the neurological state in patients suffering from traumatic SAH between the 3rd and 12th day inclusive of treatment (according to retrospective studies already carried out) and responsible for its specific morbidity linked to cerebral ischemia localized in the spasmed area manifested by a worsening of the neurological prognosis on the modified Rankin scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 or over,
* Hospitalized at the Martinique University Hospital for the treatment or monitoring of a moderate or severe TBI (Glasgow Score less than or equal to 13 at initial treatment) presenting with SAH on the cerebral CT scan,
* Patient if capable, or representative of the patient in case of incapacity, having been informed of the research, and having given free, informed and written consent,
* After an emergency inclusion procedure if the patient's representative is initially unreachable and written agreement, informed within the first 48 hours of inclusion by the representative or the patient if his neurological condition allows it,
* Be affiliated to a social security system.

Exclusion Criteria:

* Pregnant woman,
* Presence of an aneurysmal pathology known or diagnosed at initial treatment,
* History of chronic kidney failure stage 4 (creatinine clearance measured less than 30ml/min),
* Imminent death of the patient,
* Patient presenting criteria for non-admission to critical care (death expected within 48 hours, progressive fatal pathology with vital prognosis in less than 30 days, patient in palliative situation),
* Known allergy to iodized contrast products,
* Be placed under legal protection, guardianship or curatorship,
* Patient or representative who refused to allow the patient to participate in the study.

Additional Exclusion Criteria after patient's inclusion:

* Death of the patient expected within the first 48 hours,
* Minor,
* Release from hospitalization against medical advice,
* Transfer to another establishment before the 13th day of treatment (outside the Martinique University Hospital),
* Change of opinion of the patient's representative (after neurological recovery) regarding the patient's participation in research,
* Withdrawal of consent to participate in the study being supported with refusal to use the data collected until withdrawal of participation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2028-11-06 (Estimated); Study Completion 2028-12-06 (Estimated)

PRIMARY OUTCOMES:
Estimate the incidence of cerebral vasospasm (CV) with clinical impact in moderate to severeTBI patients complicated by subarachnoid hemorrhage (SAH) at Martinique University Hospital. | 42 months
  Number of incident cases of post-traumatic CV with cerebral perfusion defect observed in the event of new symptoms or neurological worsening in moderate to severe TBI between 3rd and 12th day of treatment post-traumatic in critical care during the study period.
  Incidence will be calculated by reporting the number of incident cases of traumatic CV over the total number of patients at risk (traumatic SAH) observed during the study period.

SECONDARY OUTCOMES:
Describe the characteristics of traumatic CV diagnosed in the study sample. | 42 months
  Characteristics of post-traumatic CV diagnosed in the study sample: topography (affected cerebral artery and impacted brain area)
Describe the characteristics of traumatic CV diagnosed in the study sample. | 42 months
  Characteristics of post-traumatic CV diagnosed in the study sample: time to onset
Describe the characteristics of traumatic CV diagnosed in the study sample. | 42 months
  Characteristics of post-traumatic CV diagnosed in the study sample: time to possible recurrences
Describe the characteristics of traumatic CV diagnosed in the study sample. | 42 months
  Characteristics of post-traumatic CV diagnosed in the study sample: duration of each CV episode
Analyze the risk factors for the occurrence of traumatic CV. | 42 months
  Supposed risk factors for post-traumatic CV described in the scientific literature:
  * SAH intensity (Fisher and WFNS Score, VASOGRADE Score),
  * State of consciousness at treatment (Glasgow Coma Scale at treatment),
  * Pre-existing high blood pressure,
  * Tobacco consumption,
  * Left ventricular hypertrophy,
  * Age,
  * Sex.
  The association between the presence of these factors and the occurrence of post-traumatic CV will be quantified by measures of association (odds ratio) resulting from the implementation of appropriate modeling techniques (logistic regression).
Compare the neurological morbidity at 30 days and 6 months of patients with and without post-traumatic CV in the study sample. | 42 months
  Neurological morbidity: Modified Rankin score at 1 month and 6 months after initial treatment.
  The modified Rankin Score is a disability scale used in the long-term assessment of disability linked to acute neurological pathologies (scale ranging from 0-autonomy to 6-death).
  Neurological morbidity at 1 and 6 months will be compared between patients with and without post-traumatic CV in the study sample.
Analyze the association between the worsening of the neurological prognosis 6 months after initial patient management, and the presence of a traumatic CV. | 42 months
  The association between the presence of post-traumatic CV and the worsening of the neurological prognosis (Rankin Score ≥ 4) will be quantified by the association measures (odds-ratio) resulting from the implementation of modeling techniques adequate (logistic regression).
Assess quality of life at 6 months | 42 months
  Level of quality of life at 6 months after initial treatment, assessed by the McGill questionnaire for measuring patients quality of life (McGill Quality of Life Questionnaire, revised version, MQOL-R).

CONTACTS AND LOCATIONS:
Overall Officials: Marie SABIA, PhD, Principal Investigator — University Hospital Center of Martinique
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, France

IPD SHARING:
Plan to Share IPD: No